CLINICAL TRIAL: NCT04526249
Title: Evaluation of Efficacy of the Prototype RPC (Rapid Pulse Confirmation) Device in Detecting Return of Pulsatile Flow in Patients Preparing to Separate From CPB (Cardiopulmonary Bypass)
Status: Completed | Type: Observational
Sponsor: Michael Kyle Ritchie (Other)
Collaborators: West Virginia Clinical and Translational Science Institute (Other)
Responsible Party: Sponsor-Investigator, Michael Kyle Ritchie, Primary investigator and Inventor, West Virginia University
Organization: West Virginia University (Other)
Other Study IDs: 1708690742
Record Dates: First submitted 2019-06-06; First posted 2020-08-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Circulatory Failure; Cardiac Arrest
Keywords: cardio pulmonary resuscitation; pulse detection; chest compressions
MeSH Terms: conditions — Shock; Heart Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: rapid pulse confirmation device — device used to detect pulsatile blood blood during and after cardiac arrest

SUMMARY:
Effective chest compressions are essential to survival in an arrest patient receiving CPR (cardiopulmonary resuscitation). A challenge in providing effective chest compressions is frequent interruption of compressions. A major cause of a recurrent interruption of chest compressions is pulse checks. Pulse checks are difficult to quickly and accurately perform in the AHA recommended time interval of under 10 seconds for reasons ranging from inexperience to body habitus. Unnecessarily long pulse checks often delay reinitiating chest compressions leading to a fall in perfusion pressure to the coronary arteries lowering the chances of return of spontaneous circulation (ROSC). To potentially solve the issues of evaluating the chest compression effectiveness and minimize the time interval of pulse checks, the authors have constructed a novel device that can be rapidly applied to an arresting patient and evaluate the current state of the circulatory system. The device is called the Rapid Pulse Confirmation (RPC) device. It is designed to applied over a major artery (radial, ulnar, brachial, carotid, and femoral) and detect Doppler shift of red blood cells to gauge red blood cell velocity and rate of pulsation. Feasibility testing on the device was carried out using patients requiring cardiopulmonary bypass. Arrest and return of spontaneous circulation during cardiopulmonary bypass is predictable and provided an ideal environment to test the initial performance of a device meant to detect return of spontaneous circulation. The primary working hypothesis was that there would be no significant difference in time of detection of ROSC between the arterial line catheter and the RPC device at the end of cardiopulmonary bypass. The secondary hypothesis was that there would be no difference in pulse rate reading between the arterial line catheter and the RPC device.

ELIGIBILITY:
Inclusion: 1.18 or older 2.EF >40% on pre-operative echocardiogram 3.Patient with isolated cardiac valve disease to be repaired during scheduled surgery Exclusion: 1.Redo procedure 2.Emergency procedure 3.Peripheral vascular disease 4.Previous cannulation or harvesting of radial artery 5.Arterial stents in the radial, ulnar, brachial, femoral, or carotid arteries 6.History of peripheral arterial bypass 7.History of carotid artery stenosis 8.Thoracic outlet syndrome 9.Valvular heart disease NOT being repaired day of surgery 10.Heart rhythm other than sinus prior to procedure (occasional PVC's ok) 11.Patient refusal

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled isolated open-heart valve or isolated coronary artery bypass graft surgery.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2019-01-20 (Actual); Study Completion 2019-01-20 (Actual)

PRIMARY OUTCOMES:
detection of return of spontaneous circulation by experimental device vs. indwelling arterial catheter | less than 5 minutes
  Timed in seconds

CONTACTS AND LOCATIONS:
Locations (1):
- West Virginia University Ruby Memorial Hospital, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No